CLINICAL TRIAL: NCT02123576
Title: Treatment of Type I Hepatorenal Syndrome (HRS) With Pentoxyfylline: A Placebo Controlled, Blinded Pilot Study
Brief Title: Treatment of Type I Hepatorenal Syndrome (HRS) With Pentoxyfylline
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment of study population
Sponsor: Patrick Northup, MD (Other)
Responsible Party: Sponsor-Investigator, Patrick Northup, MD, Associate Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17365
Record Dates: First submitted 2014-04-18; First posted 2014-04-25 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Hepatorenal Syndrome
Keywords: Hepatorenal syndrome; Renal failure; Pentoxyfylline; Liver transplantation; Cirrhosis
MeSH Terms: conditions — Hepatorenal Syndrome; Renal Insufficiency; Fibrosis | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Pentoxyfylline 400mg three times a day or 400mg twice a day for eGFR 10-50 and 400mg once a day for eGFR <10 for 90 days in addition to standard AMO therapy
  Interventions: Drug: Pentoxyfylline; Drug: AMO Therapy
- Placebo (Placebo Comparator): This is a standard placebo pill.
  Interventions: Drug: Placebo; Drug: AMO Therapy

INTERVENTIONS:
Drug: Pentoxyfylline
  Arms: Treatment
Drug: Placebo
  Arms: Placebo
Drug: AMO Therapy — Albumin, midodrine and octreotide therapy (standard of care for HRS)

SUMMARY:
Pentoxyfylline therapy in addition to the standard of care of albumin, midodrine and octreotide therapy is superior to the standard of care alone in the treatment of Type I hepatorenal syndrome in the first 14 days of hospitalization.

DETAILED DESCRIPTION:
Each hospitalized subject will undergo pre-dosing screening with review of his or her history and physical exam from the day of enrollment and safety assessment to ensure no contraindication to use of PTX. Type I HRS will be defined according to the criteria put forth by the American Association for the Study of Liver Disease as (1) cirrhosis with ascites; (2) serum creatinine greater than 1.5 mg/dL; (3) no improvement of serum creatinine (decrease to a level of 1.5 mg/dL or less) after at least two days with diuretic withdrawal and volume expansion with albumin; (4) absence of shock; (5) no current or recent treatment with nephrotoxic drugs; and (6) absence of parenchymal kidney disease as indicated by proteinuria >500 mg/day, microhematuria (>50 red blood cells per high power field), and/or abnormal renal ultrasonography. Baseline testing will be obtained from hospitalization records, including but not limited to chemistry panel, liver function testing, urinalysis, urine electrolytes, coagulation studies, blood cultures, chest x-ray, diagnostic paracentesis, abdominal ultrasound with Doppler.

Subjects will take either placebo three times a day or pentoxyfylline 400mg three times a day or 400mg twice a day for eGFR 10-50 and 400mg once a day for eGFR <10 for 90 days in addition to standard AMO therapy. Treatment will be continued for 14 days unless a study endpoint has been reached at which time either PTX or placebo will be stopped

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute or chronic liver disease
* Type I HRS
* Aged greater than or equal to 18
* Non-pregnant

Exclusion Criteria:

* Allergy or hypersensitivity to PTX or intolerance to methylxanthines (e.g. caffeine, theophylline)
* Concurrent use of nephrotoxic drugs
* Age less than 18
* Pregnancy
* Uncontrolled bacterial infection
* Renal parenchymal disease (e.g. acute tubular necrosis, glomerular disease, interstitial nephritis and urinary obstruction)
* Shock
* TNF alpha antagonist use
* Subject is institutionalized or a prisoner
* Recent cerebral or retinal hemorrhage (contraindication to PTX)
* Severe or poorly controlled cardiovascular disease as determined by the principal investigator to hinder the ability to adhere to study protocols

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick G Northup, MD MHS, Study Director — University of Virginia; Jonathan G Stine, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Morgan TR, McClain CJ. Pentoxifylline and alcoholic hepatitis. Gastroenterology. 2000 Dec;119(6):1787-91. doi: 10.1053/gast.2000.20826. No abstract available. PMID 11113103
- [Background] Angeli P. beta-blockers and refractory ascites in cirrhosis: the message of a team of true scientists. J Hepatol. 2011 Oct;55(4):743-4. doi: 10.1016/j.jhep.2011.02.026. Epub 2011 Mar 10. No abstract available. PMID 21396970
- [Background] Lott JP. Renal failure in cirrhosis. N Engl J Med. 2010 Jan 7;362(1):79; author reply 80-1. doi: 10.1056/NEJMc0910190. No abstract available. PMID 20054052
- [Background] Spring FA, Dalchau R, Daniels GL, Mallinson G, Judson PA, Parsons SF, Fabre JW, Anstee DJ. The Ina and Inb blood group antigens are located on a glycoprotein of 80,000 MW (the CDw44 glycoprotein) whose expression is influenced by the In(Lu) gene. Immunology. 1988 May;64(1):37-43. PMID 2454887
- [Background] Fallon E, Ehrenwald E, Nazarian GK, Smith CI. TIPS with a polytetrafluoroethylene-lined stent graft and associated haemolytic anaemia. Gut. 2008 Aug;57(8):1180-1. No abstract available. PMID 18628385

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Pentoxyfylline 400mg three times a day or 400mg twice a day for eGFR 10-50 and 400mg once a day for eGFR <10 for 90 days in addition to standard AMO therapy
  Pentoxyfylline
  AMO Therapy: Albumin, midodrine and octreotide therapy (standard of care for HRS)
- Placebo: This is a standard placebo pill.
  Placebo
  AMO Therapy: Albumin, midodrine and octreotide therapy (standard of care for HRS)
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 57 [52.4 to 61.6] | 60.8 [52.5 to 69.2] | 58.9 [52.4 to 69.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: We define this as a decrease in serum creatinine level to <1.5 mg/dL without dialysis or death
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

2. Secondary Outcome: Change in Serum Creatinine From Baseline
Time Frame: baseline and 14 days
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 6 | 6
g/dL | 0.48 [-0.49 to 1.46] | 0.03 [-0.64 to 0.70]

3. Secondary Outcome: Incidence of Treatment Failure
Description: Defined as creatinine level above baseline value after day 7, dialysis or death
Time Frame: up to day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 3 | 3

4. Secondary Outcome: Number of Participants With Combined Outcome of Treatment Success and Partial Response
Description: We define as serum creatinine level decreased by >50% from baseline but not to <1.5 mg/dL, without dialysis or HRS recurrence
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

5. Secondary Outcome: Transplant Free Survival
Time Frame: day 30 and 180
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 6 | 6
days | 80 [2 to 163] | 36 [4 to 67]

6. Secondary Outcome: Overall Survival
Description: This will be the combination of transplant free survival and those patients who received liver transplant
Time Frame: up to 1 year
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 6 | 6
days | 102 [12 to 192] | 59 [11 to 129]

ADVERSE EVENTS:
Time Frame: adverse event data was collected for up to 14 days while subject was on placebo or AMO therapy.
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 5/6 | 3/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6) | Placebo (N=6)
Discontinued intervention (General disorders) | 1 (1) | 0 (0) — nausea/vomiting

LIMITATIONS AND CAVEATS:
Small sample size due to low numbers of recruitment over a two year study period.

Inherent limitations to PTX as this medication cannot be administered through gastric feeding tube owing to it's pharmacologic properties.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT02123576/Prot_SAP_000.pdf